CLINICAL TRIAL: NCT05187078
Title: Cervical Bleeding With Cervical Stabilization During IUD Placement: Allis Clamp Versus Single-tooth Tenaculum
Brief Title: Allis Clamp Versus Single-tooth Tenaculum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Andrews (Other)
Responsible Party: Sponsor-Investigator, Brooke Andrews, Resident Physician, OB/Gyn, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-1110-P3K
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: IUD
Keywords: Cervical stabilization

STUDY DESIGN:
Who Masked: Participant
Masking Description: Physician participants were aware of assignment to utilize the single-toothed tenaculum clamp or allis clamp directly prior to IUD placement procedure. Participants were blinded to the clamp assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IUD placement with allis clamp (Experimental)
  Interventions: Procedure: Allis clamp
- IUD placement with single tooth tenaculum (Active Comparator)
  Interventions: Procedure: Single-tooth tenaculum

INTERVENTIONS:
Procedure: Allis clamp — Physicians utilized an Allis clam for cervical stabilization during IUD placement.
  Arms: IUD placement with allis clamp
Procedure: Single-tooth tenaculum — Physicians utilized a single-tooth tenaculum clam for cervical stabilization during IUD placement.
  Arms: IUD placement with single tooth tenaculum

SUMMARY:
This study aims to determine whether an Allis clamp is an effective clamp for cervical stabilization compared to a single-tooth tenaculum.

ELIGIBILITY:
Inclusion Criteria:

* Obtaining IUD

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who experienced bleeding after IUD placement | At the time of IUD insertion
  Number of patients who experienced bleeding after IUD placement with an Allis clamp or single-tooth tenaculum.

SECONDARY OUTCOMES:
IUD insertion success rate | At the time of IUD insertion
  The percentage of participants who successfully had an IUD placed with an Allis clamp or single-tooth tenaculum.
Number of interventions required for cervical clamp site bleeding hemostasis | At the time of IUD insertion
  Number of interventions required to achieve hemostasis after IUD placement with an Allis clamp or single-tooth tenaculum.
Time to hemostasis | At the time of IUD insertion
  The time in seconds required to achieve hemostasis after IUD placement with an Allis clamp or single-tooth tenaculum.
Participant reported pain | At the time of IUD insertion
  Pain reported by the participant (0-10 where a higher number indicates greater pain) at the time of IUD placement with n Allis clamp or single-tooth tenaculum.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Rone, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andrews B, Quick K, MacLeod E, Edwards K, Rone BK. Cervical bleeding with cervical stabilization during IUD placement: allis clamp versus single-tooth tenaculum, a randomized control trial. Arch Gynecol Obstet. 2023 Apr;307(4):1015-1019. doi: 10.1007/s00404-022-06784-x. Epub 2022 Dec 7. PMID 36477274